CLINICAL TRIAL: NCT00284531
Title: Use of Zenapax (Daclizumab) for the Prevention of Primary Acute Cardiac Rejection in Children and Adolescents. Ind Number: 10100
Brief Title: Use of Daclizumab for the Prevention of Allograft Rejection in Pediatric Heart Transplant Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Baylor College of Medicine (Other)
Collaborators: Roche Pharma AG (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEN122; H-18397 (Other: Baylor College of Medicine)
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Cardiac Transplantation
Keywords: cardiac transplantation; allograft rejection; anti-CD25
MeSH Terms: interventions — Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Daclizumab

SUMMARY:
This protocol is designed to obtain information on the drug levels, metabolism, and safety of daclizumab (Zenapax(R)) in children and adolescents undergoing cardiac transplantation. In addition to the drug safety and metabolism information, the number and severity of rejection episodes in patients undergoing cardiac transplantation using the standard immunosuppressive drugs plus daclizumab will be compared with patients who have previously undergone cardiac transplantation at the Baylor College of Medicine and received the same standard immunosuppressive drugs without daclizumab.

DETAILED DESCRIPTION:
Initial studies in renal and recent studies in adult cardiac transplant patients have shown Zenapax(R) to be both efficacious and safe when used in several different dosing schedules. Little data is available regarding pharmacokinetics, safety and appropriate dosing in pediatric heart transplant patients. Yet this ever-increasing group of patients presents a significant challenge for the prevention of primary rejection and the appropriate maintenance of immunosuppression. Induction of long term allograft acceptance through peripheral tolerance has been shown in animal models to be more easily induced in young animals. Once established however, allograft rejection and immunologic responses in the young are quite vigorous. This dichotomy makes young allograft recipients a particularly attractive population for the study of immune modulators targeted at preventing proliferative expansion of alloreactive T cell clones. This is precisely the mode of action of anti-IL2R monoclonal reagents such as Zenapax(R).

Although some pharmacokinetic data have been generated in adult heart transplant patients on multidrug immunosuppressive regimens including both Zenapax(R) and mycophenolate mofetil (MMF), detailed pharmacokinetic data on this combination in multidrug immunosuppressive regimens is not available for pediatric heart transplant subjects.

Objectives:

* Determination of pharmacokinetics of Zenapax(R) in pediatric patients receiving a uniform multidrug immunosuppressive regimen for primary induction.
* Determine whether there are any unusual drug interactions peculiar to the pediatric population that would require dosing modification.

Secondary objectives:

* Investigate long term effects of Zenapax(R) containing induction regimen on pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be undergoing their first cardiac allograft transplant.
* Male or female must be less than or equal to 18 years of age.
* Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to transplantation. The sensitivity must be equal to at least 50 mIU/ml. (Urine test is allowed in addition to serum test in patients where serum results are delayed.)
* Women of childbearing potential must use two reliable forms of contraception simultaneously.
* Effective contraception must be used before beginning study drug therapy, and for 4 months following discontinuation of study drug therapy.
* Patients and/or their guardians must be willing and be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

Exclusion Criteria:

* Patients with a history of hypersensitivity reactions to any of the constituents of the Zenapax(R) preparation or having had hypersensitivity reactions to human or murine immune globulin preparations in the past.
* Women lactating, pregnant or of childbearing potential not using, or who are unwilling to use two reliable forms of contraception simultaneously during the study
* History of a psychological illness or condition which would interfere with the patient's ability to understand the requirements of the study
* White blood count < 2500/mm^3, platelets < 50,000 /mm^3 or hemoglobin < 6 g/dL.
* HIV-1 infection or the presence of positive hepatitis B surface antigen (HBsAg) or chronic hepatitis C.
* Active peptic ulcer disease
* Severe diarrhea or other gastrointestinal disorders which might interfere with the ability to absorb oral medication
* Malignancies within the past 5 years, excluding skin carcinomas (basal or squamous cell) that have been adequately treated
* Patients who have received within the past 30 days or require concomitant treatment with other investigational drugs or immunosuppressive medications that are prohibited for this study
* Inability to start microemulsion form of cyclosporine within 72 hours

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2003-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Drug levels at scheduled time points
Receptor saturation at scheduled time points
Number of rejection episodes in 1 year

SECONDARY OUTCOMES:
Changes in T cell subsets over observation period
Numbers of bacterial and opportunistic infections
Evidence for autoimmune disease over observation period

CONTACTS AND LOCATIONS:
Overall Officials: Howard M Rosenblatt, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States